CLINICAL TRIAL: NCT06310213
Title: Non-Invasive Pressure Monitor for Neonates & Infants at Risk of Developing Hydrocephalus
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jignesh Tailor, Assistant Professor of Neurological Surgery, Indiana University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 17368
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Hydrocephalus in Infants

STUDY DESIGN:
Intervention Model Description: Aim 1: Comparison of neonates and infants with hydrocephalus and without Aim 2: Using smart soft contact lens (SSCL) for pre- and post-operative measurements on neonates and/or infants managed operatively (shunt placement) Aim 3: Direct validation by comparing SSCL to external ventricular drain (EVD) intracranial pressure (ICP) monitoring Aim 4: Using SSCL for pre- and post- reservoir tap measurements on neonates and/or infants managed operatively (reservoir placement) Aim 1: 10 patients per arm, two arms Aim 2: 5-10 patients, one arm Aim 3: 5-10 patients, one arm Aim 4: 5-10 patients, one arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (5):
- Aim 1 Control (Active Comparator): Intervention at single time point not to interfere with standard of care procedures
  Interventions: Device: Non-Invasive Pressure Monitor
- Aim 1 Hydrocephalus (Experimental): Intervention at single time point during standard of care hydrocephalus evaluation (anterior fontanelle assessment and measurement of head circumference), unless further assigned to supplemental arm following standard of care surgical procedure
  Interventions: Device: Non-Invasive Pressure Monitor
- Aim 2 Hydrocephalus, Shunt surgery (Experimental): Intervention pre- and post-operatively
  Interventions: Device: Non-Invasive Pressure Monitor
- Aim 3 Hydrocephalus, EVD ICP monitor (Experimental): Intervention during standard of care monitoring of EVD ICP reading(s)/hydrocephalus evaluation (anterior fontanelle assessment and measurement of head circumference)
  Interventions: Device: Non-Invasive Pressure Monitor
- Aim 4 Hydrocephalus, Reservoir surgery (Experimental): Intervention pre- and post- ventricular reservoir tap(s)
  Interventions: Device: Non-Invasive Pressure Monitor

INTERVENTIONS:
Device: Non-Invasive Pressure Monitor — Modified smart soft contact lens and cap with reader coil

SUMMARY:
The goal of this clinical trial is to test a modified smart soft contact lens in neonates and infants at risk of developing hydrocephalus. The main questions it aims to answer are:

* Can the device distinguish between intracranial pressure variations in neonates and infants diagnosed with hydrocephalus and those without
* Can the device compare pressure dynamics between pre- and post-operative periods in neonates and infants who undergo surgical treatments Participants will undergo standard of care evaluations for hydrocephalus (anterior fontanelle assessment and head circumference measurement) and wear the device during standard of care evaluation; pre- and post- ventricular reservoir taps, as applicable; and/or pre- and post-operatively, as applicable.

ELIGIBILITY:
Inclusion Criteria:

* Being monitored for hydrocephalus, or healthy controls

Exclusion Criteria:

* Known hypersensitivity to materials used in the contact lens and/or adhesive
* Open/closed wounds at/near the anterior fontanelle
* Anterior fontanelle is closed
* Other conditions deemed relevant by the medical team

Ages: 0 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of modified smart soft contact lens evaluation of external intracranial pressure at single time point (Aim 1) | Day 1, continuously measured for up to 4 hours
  ICP readings from the device will be compared to standard of care assessments and measurements in healthy control patients and hydrocephalus patients
Efficacy of modified smart soft contact lens evaluation of external intracranial pressure before and after shunt surgery (Aim 2) | Continuously measured for up to 4 hours prior to shunt surgery and continuously measured for up to 4 hours after shunt surgery
  ICP readings from the device will be compared to standard of care assessments and measurements in patients undergoing shunt insertion
Efficacy of modified smart soft contact lens evaluation of external intracranial pressure during hydrocephalus evaluation (Aim 3) | Continuously measured for up to 4 hours while EVD/ICP monitoring is in place
  ICP readings from the device will be compared to standard of care assessments and measurements in patients with an EVD/ICP monitor
Efficacy of modified smart soft contact lens evaluation of external intracranial pressure before and after reservoir taps (Aim 4) | Continuously measured for up to 4 hours prior to reservoir tapping and continuously measured for up to 4 hours after reservoir tapping
  ICP readings from the device will be compared to standard of care assessments and measurements in patients with a reservoir, pre- and post-tap

CONTACTS AND LOCATIONS:
Overall Officials: Jignesh Tailor, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No